CLINICAL TRIAL: NCT02234895
Title: Combined Medial and Lateral Orthotics for the Treatment of Knee Osteoarthritis
Brief Title: Shoe Orthotics for Improvement of Biomechanics and Symptoms of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Pedorthic Research Foundation of Canada (Unknown); Kintec Footlabs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H14-01313
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee; biomechanics; treatment; symptoms
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lateral wedge plus medial arch support (Experimental): The lateral wedge plus medial support orthotic will be custom-made and designed using a 3D volumetric cast of the foot with the participant's foot in a subtalar joint neutral position. The cast will be balanced so that it rests in a neutral position then smoothed to address any irregularities and to allow for soft tissue splay. Polypropylene sheets of 3mm or 4mm thickness will be vacuum formed or milled directly to produce a ¾ length shell. An ethyl-vinyl-acetone (EVA) lateral post in the heel and forefoot of 5 degrees will be incorporated into the orthotic. The orthotic will be finished with a neoprene cover for improved comfort and patient compliance.
  Interventions: Device: Lateral wedge plus medial arch support
- Lateral wedge (Experimental): The lateral wedge only orthotic will be constructed of EVA, made to full length of the subject's footwear and incorporate a 5 degree posting. The wedge will be finished with a neoprene cover for improved comfort and patient compliance.
  Interventions: Device: Lateral wedge

INTERVENTIONS:
Device: Lateral wedge — This will be a randomized cross-over study where all participants will receive both orthoses over a six month period. Each intervention will last two months, separated by a two month washout period of no orthotics wear, and will be preceded and followed by a laboratory-based gait and pain assessment. Two months has been chosen as the ideal time frame to ensure maximum participant adherence, to observe clinically meaningful changes in symptoms, and to minimize degradation of the insoles.
  Arms: Lateral wedge
Device: Lateral wedge plus medial arch support — This will be a randomized cross-over study where all participants will receive both orthoses over a six month period. Each intervention will last two months, separated by a two month washout period of no orthotics wear, and will be preceded and followed by a laboratory-based gait and pain assessment. Two months has been chosen as the ideal time frame to ensure maximum participant adherence, to observe clinically meaningful changes in symptoms, and to minimize degradation of the insoles.
  Arms: Lateral wedge plus medial arch support

SUMMARY:
Knee osteoarthritis (OA) is a widespread problem in Canada, leading to decreased quality of life and increased economic burden. Current research has focused on expensive, invasive treatments, whereas inexpensive conservative treatments have received less attention. One such treatment is the use of orthotics to reduce pain and increase function in people with knee OA. Currently, clinical practice guidelines for the use of orthotics are vague and contradictory, and could benefit from more research taking into account foot posture. This study aims to compare the use of two orthotics designs in people with knee OA.

ELIGIBILITY:
Inclusion Criteria:

i) age 50 - 80 years (to meet the American College of Rheumatology clinical definition of OA)

ii) medial tibiofemoral OA, defined as medial knee pain on most days of the past month and evidence on radiographs of a definite osteophyte in the medial tibiofemoral compartment

iii) pronated feet, defined as a foot posture index that is 0.5 standard deviations above the reported population mean.

Exclusion Criteria:

i) low pain score on a numerical rating scale of pain (average knee pain on walking ≤3 out of 10 over previous week) to allow detection of treatment response

ii) knee surgery or intra-articular corticosteroid injection within the previous six months

iii) current or recent (within 4 weeks) oral corticosteroid use

iv) any muscular, joint or neurological condition affecting lower limb within the past 6 months

v) ankle/foot pathology or pain that precludes the use of orthotics

vi) current use of foot orthotics

vii) use of footwear unable to accommodate an orthotic

viii) unable to walk without a gait aid

ix) inability to speak English or have a family member present to translate (required for the validity of the questionnaires)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in knee joint load during walking: knee adduction moment | Baseline and 2 months
  Participants will undergo three-dimensional gait analysis. This will be performed barefoot with and without the orthotics (conditions tested in a random order). Kinematic and kinetic data will be collected synchronously using high-speed digital cameras and floor-mounted force platforms. Participants will be instructed to walk at a self-selected walking speed measured using photoelectric timing gates and placed along the walkway two metres on either side of the force platforms (note that walking speed during follow-up assessments will be kept similar (+/- 5%) to that chosen by each participant at baseline). A total of five trials will be collected.
  The primary loading variable will be the KAM impulse - defined as the area under the KAM curve. Rather than a single peak value, the KAM impulse is more reflective of load experienced over the duration of stance and reflects the cumulative loading experienced at the knee during walking.
Change in Knee Pain | Baseline and 2 Months
  The WOMAC is a disease-specific questionnaire that quantifies self-reported joint pain, joint stiffness, and physical function. It is a valid, reliable, and responsive outcome measure that is recommended for use in osteoarthritis clinical trials.

SECONDARY OUTCOMES:
Change in Self-Reported Physical Function | Baseline and 2 Months
  The physical function subscale (17 questions) on the WOMAC will be used.
Change in Foot Pain | Baseline and 2 Months
  Participants will rate their perceived foot function and pain using the Foot Function Index (revised - short form). This is a self-report questionnaire which consists of 34 items and provides the ability to quantify aspects of pain, disability and activity limitation. Such assessment of pain has been widely used and is a valid and reliable method in clinical research studies

OTHER OUTCOMES:
Participant perceived response to treatment | 2 Months
  At follow-up for each orthotic, participants will rate overall perceived change in pain and physical function (vs. baseline) on an ordinal scale (1-much worse, 2-slightly worse, 3-same, 4-slightly better, 5-much better). This will be dichotomized into 'improvement' (4 and 5) or 'no improvement'

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Hunt, PhD, PT, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia; University Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Hunt MA, Takacs J, Krowchuk NM, Hatfield GL, Hinman RS, Chang R. Lateral wedges with and without custom arch support for people with medial knee osteoarthritis and pronated feet: an exploratory randomized crossover study. J Foot Ankle Res. 2017 May 2;10:20. doi: 10.1186/s13047-017-0201-x. eCollection 2017. PMID 28473871